CLINICAL TRIAL: NCT06738004
Title: A National Multi-centre Prospective Audit of Unplanned Surgical and Endoscopic Interventions in Patients Who Have Undergone Bariatric Surgery in the UK or Abroad
Brief Title: National Emergency Bariatric Surgery Audit
Acronym: NEBSA
Status: Recruiting | Type: Observational
Sponsor: Bedfordshire Hospitals NHS Foundation Trust (Other)
Collaborators: Alan Askari (Unknown); Aruna Munasinghe (Unknown); Omer Al-taan (Unknown); Fahad Iqbal (Unknown); Dimitri Pournaras (Unknown); Matthew Lee (Unknown); Roxanna Zakeri (Unknown); Marianne Hollyman (Unknown)
Responsible Party: Principal Investigator, Mohamed Aly, Consultant Upper GI and General Surgeon, Bedfordshire Hospitals NHS Foundation Trust
Other Study IDs: NEBSA1
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Bariatric Surgery; Postoperative Complications; Emergencies; Surgical Procedures, Operative; Outcome Assessment (Health Care); Quality Improvement; Morbidity; Mortality
Keywords: Bariatric surgery; Emergency complications; National audit; Surgical outcomes; Management strategies; United Kingdom; Patient safety; Quality improvement; Morbidity and mortality; Postoperative complications
MeSH Terms: conditions — Postoperative Complications; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to investigate the incidence, management, and outcomes of complications following bariatric surgery in patients in the United Kingdom. The main questions it aims to answer are:

* What is the prevalence of unplanned interventions due to complications following bariatric surgery in the UK?
* What are the current practices for managing these complications, and how do they impact patient outcomes?

Participants will:

Be identified from hospitals treating patients presenting with complications following bariatric surgery.

Have their data collected regarding demographics, surgical history, complications, treatments, and outcomes.

Researchers will compare different management strategies and their impact on patient outcomes, with the aim of identifying best practices to improve emergency bariatric care and factors leading to patients attending as an emergency.

DETAILED DESCRIPTION:
The National Emergency Bariatric Surgery Audit (NEBSA) is an observational study aimed at investigating the incidence, management, and outcomes of complications following bariatric surgery in the United Kingdom. The detailed description of the protocol includes the following components:

Patient Recruitment and Data Collection:

Patients will be identified in hospitals across the UK where they present for an unplanned intervention to treat a complication related to or following bariatric surgery.

Data on demographics, surgical history, site and type of index bariatric surgery, comorbidities, complications, treatments, and outcomes will be collected through a combination of electronic health records and manual data extraction.

Quality Assurance Plan:

Data checks will be performed to ensure range, completeness and consistency with other data fields in the registry.

Data entry is restricted in most fields of the data form to ensure conformity of the entries and facilitate analysis.

Sample Size Assessment:

This is a prospective observational study, so a sample size assessment is not required. Data collection will continue for a six month period per centre then analysed to report any statistically significant findings.

Plan for Missing Data:

Missing data is reported back to the collaborating sites to complete.

Statistical Analysis Plan:

The Shapiro-Wilk test will be used to check variables for Gaussian distribution. Basic demographics will be presented as absolute numbers of participants with the respective percentage per group or as parameter mean and standard deviation or median and range, depending on distribution. For comparisons of interval-scaled variables, unpaired t tests will be performed. Nonparametric between-group testing will be undertaken with 2-tailed Mann-Whitney U tests. Additionally, the chi-square test or Fisher exact test will be applied to nominal scale data. Multivariable linear regression be performed for differences among baseline demographics. Analyses will be performed in RStudio with significance defined with p < 0.05.

The NEBSA will provide valuable insights into the prevalence, management, and outcomes of complications following bariatric surgery in the UK. By comparing different management strategies and their impact on patient outcomes, this study aims to identify best practices for emergency bariatric care, ultimately improving patient outcomes and overall healthcare quality. Another important aim is analysing the effect of patient demographics, and engagement with NHS specialised weight loss services on the choice of route for bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Admissions from i) the emergency department, clinic, urgent care or primary care to the bariatric surgical team as an emergency; ii) from an inpatient team as an urgent referral; iii) a return to theatre following an elective bariatric procedure; iv) another hospital via patient transfer to a specialised unit.
* Participants undergoing any intervention or procedure to treat or diagnose bariatric complications, (e.g., OGDs, interventional radiology, surgery, supplemental enteral or parenteral nutrition).

Exclusion Criteria:

* age <18 years old
* have a length of stay <24 hrs.
* initial diagnosis of BSE is changed or if their readmission is found to be unrelated to previous bariatric surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted from these locations i) the emergency department, clinic, urgent care or primary care to the bariatric surgical team as an emergency; ii) from an inpatient team as an urgent referral; iii) a return to theatre following an elective bariatric procedure; iv) another hospital via patient transfer to a specialised unit,with the intent to treat or diagnose complications of bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2025-12-09 (Estimated); Study Completion 2025-12-09 (Estimated)

PRIMARY OUTCOMES:
30-day mortality | up to 30 days from procedure or admission
  Time in days
Inpatient length of stay | Up to 100 weeks from admission
  Time in days
Clavien-Dindo Classification of Complications | through study completion, an average of 1 year
  Severity of complication

SECONDARY OUTCOMES:
Frequency and rate of nutritional support | through study completion, an average of 1 year
  Rate of enteral, or parenteral nutritional support
Frequency and type of interventional radiology | through study completion, an average of 1 year
  Need for drains or other radiological procedures
Frequency and type of surgery, diagnostic or therapeutic procedures | through study completion, an average of 15 years post-op from index surgery
  Description of the type of procedure or intervention required to treat or diagnose complications following bariatric surgery
Frequency of admission to critical care units | through study completion, an average of 1 year
  Identify need for critical care
Engagement with NHS specialised weight management services | through study completion, an average of 10 years prior to admission
  Identify engagement with NHS services for bariatric surgery
Site and time of index bariatric surgery | Time from index surgery to admission
  Whether patient had surgery at the admitting hospital, other site in the UK or abroad

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Aly, FRCS, Principal Investigator — The Hillingdon Hospitals NHS Foundation Trust
Locations (1):
- Luton and Dunstable Hospital, Luton, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided